CLINICAL TRIAL: NCT01284465
Title: A Comprehensive Approach to Type 2 Diabetes Self-management for Low-income Women
Brief Title: Type 2 Diabetes Self-management Intervention for Low-income Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meharry Medical College (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Sylvie Akohoue, Assistant Professor, Meharry Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 081204AAH231 26; U54RR026140-01 (NIH)
Record Dates: First submitted 2011-01-25; First posted 2011-01-27 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes self-management; Minority women; Barriers to diabetes self-management
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Educational Status; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Education and patient liaison combination
  Interventions: Behavioral: Education and patient liaison combination
- Control group (Experimental): Education only
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: Education and patient liaison combination — Group education sessions with Patient liaison using ecological momentary assessment principles
  Other Names: Type 2 diabetes self-management; Low-income women; Barriers to diabetes self-care
  Arms: Intervention group
Behavioral: Control group — Group education sessions at baseline, 3 and 6 months
  Other Names: Type 2 diabetes self-management; Low-income women; Barriers to diabetes self-care
  Arms: Control group

SUMMARY:
The purpose of this study is to assess the extent to which a culturally appropriate, self-management intervention that combines patient education with a patient outreach liaison strategy improves outcomes associated with type-2 diabetes among low-income diabetic women.

DETAILED DESCRIPTION:
In recent years, the prevalence of diabetes has significantly increased among women and because of the expected fast growth rate of minority populations, the number of women in these groups who will be diagnosed with diabetes is also expected to increase significantly over the coming years. Among women from minority groups diabetes is the fourth leading cause of death while it is the seventh among non-Hispanic White females. Non-compliance to diabetes self-care is a major concern for type 2 diabetic women of racial/ethnic groups because of the existing socio-economic and environmental barriers. Often, these women live in poverty; have less than a high school education as well as language barriers and inadequate health literacy, which further place them at risk for complications, and the daily activities of diabetes self-care are implemented within the context of family responsibilities and patient's priorities.

This study is a 12-month randomized controlled trial designed to compare a lifestyle intervention group (combination group) and a control group (education only group). Participants assigned to either group will receive three group education sessions (baseline, 3 and 6 months) with an emphasis on self-management.

ELIGIBILITY:
Inclusion Criteria:

1. Low-income women ages 21 and older; With type 2 diabetes ( fasting plasma glucose > 126 mg/dl);
2. At risk of developing diabetes related complications (treatments goals from The American Diabetes Association Standards of medical care) as defined by:

   * HbA1c >8.0 %
   * Any of the metabolic clusters such as Pre-prandial plasma glucose > 130 mg/dl; Obesity (BMI >25 kg/m2, or waist circumference >88 cm (>35 in); Hypertension (Systolic >130 and Diastolic > 80 mmHg); Hyperlipidemia (Triglycerides >150 mg/dL; HDL<50 mg/dL; LDL >100 mg/dL)

Exclusion Criteria:

* Participants will be excluded if they are currently pregnant, have conditions (i.e., end stage diagnosis) or behaviors likely to affect conduct of the trial, and unwilling to accept treatment assignment by randomization.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2011-01; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
HbA1c | baseline, 6 and 12 months
  glycosylated hemoglobin

SECONDARY OUTCOMES:
Risk factors for co-morbidity and daily self-management behaviors | baseline, 3, 6, 9 and 12 months
  1. -Risk factors for co-morbidity:
  2. -Daily self-management behaviors

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie A Akohoue, PhD, Principal Investigator — Meharry Medical College
Locations (1):
- Meharry medical College, Nashville, Tennessee, United States